CLINICAL TRIAL: NCT05968053
Title: Presence of Microplastics and Nanoplastics in Neurosurgery Patients
Brief Title: Detection of Microplastics and Nanoplastics in Neurosurgery Patients (DT-MiNi)
Acronym: DT-MiNi
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Xiaolin Chen, MD, Director, Beijing Tiantan Hospital
Other Study IDs: DT-MiNi
Record Dates: First submitted 2023-07-06; First posted 2023-08-01 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Carotid Artery Stenosis; Glioma; Intracranial Aneurysm; Intracranial Hemorrhages; Brain Tumor
Keywords: microplastics; nanoplastics; Intracranial Aneurysm; brain tumor; Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis; Glioma; Intracranial Aneurysm; Intracranial Hemorrhages; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: biological samples analysis — biological samples analysis

SUMMARY:
Plastic particles are a ubiquitous pollutant in the living environment and food chain, so far, plenty of studies have reported the internal exposure of microplastics and nanoplastics in human tissues and enclosed body fluids.

Neurosurgery is the only department that can open the skull. In addition to blood and cerebrospinal fluid, there are brain tissue and tumors in the presence of lesions. Whether any of these microplastics and nanoplastics are present remains a mystery. This prospective observational study will harvest biological samples of neurosurgery patients.

The objective of this research is to be able to detect microplastics and nanoplastics on blood and operation samples of neurosurgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Any type of neurosurgery

Exclusion Criteria:

·refusal of the patient to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included patients age 18-80 years with any types of neurosurgery Excluded patients refuse to participate
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
microplastics | baseline, intraoperative
  Detection of microplastics in human brain tissue and the blood undergoing neurosurgery
nanoplastics | baseline, intraoperative
  Detection of nanoplastics in human brain tissue and the blood undergoing neurosurgery

CONTACTS AND LOCATIONS:
Overall Officials: Runting Li, MD, Principal Investigator — Beijing Tiantan Hospital; Yitong Jia, MD, Principal Investigator — Beijing Tiantan Hospital; Ke Wang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided